CLINICAL TRIAL: NCT00931619
Title: GABA/Glutamate Balance in Temporal Lobe Epilepsy With and Without Major Depression
Status: Completed | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 090182; 09-N-0182
Record Dates: First submitted 2009-07-01; First posted 2009-07-02 (Estimated); Last update posted 2019-12-17 (Actual); Status verified 2013-04-02

CONDITIONS: Epilepsy; Epilepsy, Temporal Lobe; Depression; Depressive Disorder, Major
Keywords: Fluorine-18 Fluorodeoxyglucose; Epilepsy; Epileptic Focus; Temporal Lobe Epilepsy; Depression; Major Depressive Disorder; Healthy Volunteer; HV
MeSH Terms: conditions — Epilepsy; Epilepsy, Temporal Lobe; Depression; Depressive Disorder, Major

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
Objective: To study the relative balance of GABA (A) binding potential and glutamate utilization in subjects with localization-related epilepsy with and without depression, subjects with major depressive disorder alone, and in subjects with generalized epilepsy (expected not to have significant comorbid depression). Pilot data shows that GABA(A) binding potential and glutamate utilization are tightly coupled in healthy subjects particularly in the mesial temporal lobe. We hypothesize that subjects with epilepsy will not exhibit the same degree of coupling, and that subjects with both epilepsy and depression will exhibit an even more pronounced decoupling.

Study Population: Subjects aged 18-55 with localization-related epilepsy with and without depression, subjects with generalized epilepsy, subjects with major depressive disorder (MDD) alone, and healthy controls.

Design: This is a neuroimaging study, using positron emission tomography (PET) with [11C]flumazenil, to measure GABA(A) binding potential, and [18F]fluorodeoxyglucose, to measure glucose utilization (reflective of neuronal glutamate release) Magnetic resonance spectroscopy (MRS), will be used to measure GABA and glutamate in the mesial temporal cortex, and corroborate the PET results. Structural magnetic resonance images (MRI) will be obtained for MRS localization and partial volume correction of PET images.

Outcome measures: The binding potential of GABA(A), the regional rate of glucose metabolism, and the levels of GABA and glutamate as measured by MRS. Patients will be stratified by seizure type and depression ratings.

...

DETAILED DESCRIPTION:
Objective: To study the relative balance of GABA (A) binding potential and glutamate utilization in subjects with localization-related epilepsy with and without depression, subjects with major depressive disorder alone, and in subjects with generalized epilepsy (expected not to have significant comorbid depression). Pilot data shows that GABA(A) binding potential and glutamate utilization are tightly coupled in healthy subjects, particularly in the mesial temporal lobe. We hypothesize that subjects with epilepsy will not exhibit the same degree of coupling, and that subjects with both epilepsy and depression will exhibit an even more pronounced decoupling.

Study Population: Subjects aged 18-55 with localization-related epilepsy without clinically significant depression, subjects with generalized epilepsy, and healthy controls.

Design: This is a neuroimaging study, using positron emission tomography (PET) with [11C]flumazenil, to measure GABA(A) binding potential, and [18F]fluorodeoxyglucose, to measure glucose utilization (reflective of neuronal glutamate release). Magnetic resonance spectroscopy (MRS) will be used to measure GABA and glutamate in the mesial temporal cortex and corroborate the PET results. Structural magnetic resonance images (MRI) will be obtained for MRS localization and partial volume correction of PET images.

Outcome measures: The binding potential of GABA(A), the regional rate of glucose metabolism, and the levels of GABA and glutamate as measured by MRS. Patients will be stratified by seizure type.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Male and female subjects aged between 18 and 55 years
* Epileptic patients must have clinically documented partial seizures, in either the left or right temporal lobe, or generalized seizures with consistent EEG evidence as defined by the 1981 International Classification of Epileptic Seizures, refractory to standard antiepileptic treatment for at least one year. This criterion will be established by preliminary screening in the NINDS CES outpatient clinic, and, where previous studies are not adequate, by inpatient video-EEG monitoring.
* All subjects with epilepsy must exhibit seizures not adequately controlled by medication alone, despite adequate trials of multiple agents.

Subjects with epilepsy must currently be taking an AED which exerts its primary method of action on a system other than GABA. Examples include sodium or calcium channel blockers (phenytoin, carbamazepine, oxcarbazepine, lamotrigine, zonisamide, and ethosuximide), drugs that bind to SV2A sites (levetiracetam), or drugs which bind to the alpha2delta subunit of calcium channels (gabapentin and pregbalin). Patients on AEDs that have direct effects on GABA and glutamate (vigabatrin, phenobarbital, benzodiazepines, tiagabine) will be excluded. No subject s medication will be changed for the purpose of inclusion in this study.

* Patients with TLE and depression must currently meet DSM-IV criteria for the category "Mood disorder due to epilepsy" (293.83), and the subtype "with Major Depressive-Like Episode", 296.2 Major Depressive Disorder, Single Episode, or 296.3 Major Depressive Disorder, Recurrent, indicating that subjects meet diagnostic criteria for a major depressive episode.
* Patients with MDD alone must currently meet DSM-IV criteria for Major Depressive Disorder, and also have either a family history of mood disorders, or a history of multiple major depressive episodes.
* Healthy control subjects who do not meet criteria for any DSM-IV axis I psychiatric disorder, and have no family history (in first degree relatives) of a mood or anxiety disorder will also be recruited.
* Subjects must be able to give written informed consent prior to participation in this study.

EXCLUSION CRITERIA:

* Subjects with major medical or neurological disorders (besides TLE or generalized epileptiform disorder) expected to influence cerebral blood flow or morphology
* Subjects with epilepsy taking any medications (other than antiepileptic drugs) that may affect cerebral blood flow, GABA or glutamate neurotransmission, or metabolism.
* Subjects with epilepsy taking AED s known to exert direct effects on GABA or glutamate.
* Subjects with epilepsy with depression who have taken anti-depressant drugs within 2 weeks of the study (4 weeks for fluoxetine)
* Medically healthy depressed subjects who have taken any drugs, including anti-depressants, expected to influence cerebral blood flow, metabolism, or morphology within 2 weeks of the study (4 weeks for fluoxetine)
* Healthy subjects who are taking any medications expected to influence cerebral blood flow, metabolism, or morphology.
* Healthy subjects must be free from a personal history of seizure disorders
* In order to exclude subjects at-risk for the development of a mood disorder, healthy control subjects must be free from either a personal or family history (first-degree relatives) of Axis I psychiatric disorders
* Subjects with a history of drug or alcohol abuse within one year, or a lifetime history of alcohol or drug dependence (DSM-IV criteria). Subjects who consume an excessive amount of alcohol (more than 7 drinks per week for women, more than 14 drinks per week for men) will also be excluded.
* Subjects with structural lesions visible on MRI, excluding mesial temporal sclerosis
* Subjects with suicidal ideation, or a past history of suicide attempts
* Subjects with psychotic symptoms
* Subjects in whom MRI is contraindicated
* Female subjects who are lactating or pregnant
* Subjects with an IQ of less than 80 will be excluded from the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 29 (Actual)
Dates: Start 2009-06-29; Study Completion 2013-04-02

PRIMARY OUTCOMES:
The primary outcome measures will include GABA(A) binding potential and regional glucose metabolic rate as measured by PET, and GABA and glutamate levels as measured by MRS.

SECONDARY OUTCOMES:
Secondary outcome measures will include brain structure on MRI, blood oxygenation level dependent contrast in functional resting state scans, genetic data, and scores on depression rating scales.

CONTACTS AND LOCATIONS:
Overall Officials: William H Theodore, M.D., Principal Investigator — National Institute of Neurological Disorders and Stroke (NINDS)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Baker GA, Nashef L, van Hout BA. Current issues in the management of epilepsy: the impact of frequent seizures on cost of illness, quality of life, and mortality. Epilepsia. 1997;38 Suppl 1:S1-8. doi: 10.1111/j.1528-1157.1997.tb04511.x. PMID 9092951
- [Background] Hanai T. Quality of life in children with epilepsy. Epilepsia. 1996;37 Suppl 3:28-32. doi: 10.1111/j.1528-1157.1996.tb01816.x. PMID 8681908
- [Background] Leidy NK, Elixhauser A, Vickrey B, Means E, Willian MK. Seizure frequency and the health-related quality of life of adults with epilepsy. Neurology. 1999 Jul 13;53(1):162-6. doi: 10.1212/wnl.53.1.162. PMID 10408553
- [Derived] Nugent AC, Martinez A, D'Alfonso A, Zarate CA, Theodore WH. The relationship between glucose metabolism, resting-state fMRI BOLD signal, and GABAA-binding potential: a preliminary study in healthy subjects and those with temporal lobe epilepsy. J Cereb Blood Flow Metab. 2015 Mar 31;35(4):583-91. doi: 10.1038/jcbfm.2014.228. PMID 25564232